CLINICAL TRIAL: NCT02551510
Title: Open, Randomized, Controlled Non-inferiority Trial to Compare Synthetic Tissue Adhesive and Skin Suture After Port Catheter Implantation With Reference to Cosmetic Result and Economy of Time at Equal Risk for Wound Infection
Brief Title: Comparison of Skin Adhesive to Subcuticular Suture Wound Closure After Port Placement
Acronym: PWC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Collaborators: Aesculap AG (Industry)
Responsible Party: Principal Investigator, Ulf Teichgräber, Prof. Dr. med., Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4164-07/14
Record Dates: First submitted 2015-08-17; First posted 2015-09-16 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Wound Closure After Port Catheter Implantation
Keywords: Skin Adhesive; Suture; Port Incisions
MeSH Terms: interventions — Sutures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Suture (Active Comparator): Skin incision closure with standard subcuticular technique
  Interventions: Procedure: Suture
- Experimental: Histoacryl® (Active Comparator): Skin incision closure with topic skin adhesive Histoacryl®
  Interventions: Device: Experimental: Histoacryl®

INTERVENTIONS:
Procedure: Suture — Skin incision closure with standard subcuticular technique
  Arms: Suture
Device: Experimental: Histoacryl® — Skin incision closure with topic skin adhesive Histoacryl® Flexible (n-Butyl-2-Cyanoacrylate Monomer)
  Arms: Experimental: Histoacryl®

SUMMARY:
Port Wound Closure compares synthetic tissue adhesives with seam for cutaneous wound closure to port plant in terms of cosmetic results and time savings at comparable risk for wound infection.

DETAILED DESCRIPTION:
Study patients who undergo a subcutaneous venous port implant procedure are randomized into control group (conventional sutures) or into interventional group (synthetic tissue adhesive). The intervention time is documented. Follow-up visit is performed 8 weeks after port implantation. It includes a photo documentation, quality of life questionnaire (EQ5D) and pain scala questionnaire (POSAS) by patient and by 3 independent observers as well as the documentation of complications.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication for port catheter implantation because of chemotherapy or parenteral nutrition

Exclusion Criteria:

* Children and adolescents < 18 years
* Thrombocytes < 50/nl
* PTT <50%
* INR >1.5
* Systemic or local infection of the interventional location
* Known allergy to used material
* Known allergy to Histoacryl, Cyanoacrylate, D&C Violett or Formaldehyd
* General contraindication of port catheter implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Cosmetic outcome after wound healing | 8 weeks
  Wound assessment by 3 independent evaluators (surgeons) and patient himself based on photo documentation
Cosmetic outcome after wound healing | 8 weeks
  Patient and observer scar assessment scale (POSAS)
Cosmetic outcome after wound healing | 8 weeks
  Life quality questionnaire EQ5D

SECONDARY OUTCOMES:
Infection rate | 8 weeks
  Assessment of adverse events through AE documentation based on the adverse impact of surgical site infections (German: CDC Kriterien)
Economy of time for wound closure | 10 minutes
  Time measurement by stopwatch and exact documentation of intervention time of subcutaneous suture and skin closure time

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Jena, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Witting S, Ingwersen M, Lehmann T, Aschenbach R, Eckardt N, Zanow J, Fahrner R, Lotze S, Friedel R, Lenz M, Schmidt C, Miguel D, Ludriksone L, Teichgraber U. Wound Closure After Port Implantation-A Randomized Controlled Trial Comparing Tissue Adhesive and Intracutaneous Suturing. Dtsch Arztebl Int. 2021 Nov 5;118(44):749-755. doi: 10.3238/arztebl.m2021.0324. PMID 34615593